CLINICAL TRIAL: NCT00155051
Title: Progestin Treatment for Endometrial Stromal Cells in Adenomyosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361700762; NTUH.94S72
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2004-06

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Long term treatment of progestin has been demonstrated to have an inhibitory effect on endometrial angiogenesis and the proliferation of endometrial stromal cells. As a result, progestin is now widely employed in the treatment of endometrial cancer, endometrial hyperplasia, and dysfunction uterine bleeding. In the treatment of adenomyosis, however, the beneficial effect of progestin was limited. It might imply that the behavior of endometrial cells in women with adenomyosis is different from that in women without adenomyosis.

Our previous study revealed that the expression of killer inhibitory receptors (KIRs) on NK cells was decreased in eutopic endometrium in women with adenomyosis. It may be a compensatory effect in which the NK cytotoxicity is activated in order to wipe out the abnormal endometrial cells that might go out of the eutopic site of endometrium. It implies that the formation of adenomyosis might be due to "abnormal" endometrial tissues, but not the aberrant local immunological dysfunction in myometrium. This finding is compatible with previous reports in which eutopic endometrium obtained from women with endometriosis or adenomyosis was found to behave differently from endometrium in unaffected women.

In this study, we try to collect endometrial tissues from women with and without adenomyosis, and then purify the endometrial stromal cells from endometrium. The endometrial stromal cells are cultured for 8 days with the supplement of medroxyprogesterone (MPA) or danazol. Quantification of IL-6 and IL-8 mRNA in endometrial cells, and the concentrations of IL-6 and IL-8 in cultured media will be done with real time RT-PCR and ELISA respectively. The expression of different cytokines of endometrial cells in response to progestin might be further elucidated after our experiment.

DETAILED DESCRIPTION:
Eutopic endometrium was obtained and separated into single endometrial stromal cell (ESC) in women with adenomyosis (study group) and without adenomyosis (control group).

After becoming pre-confluent (covering 80% of the culture well), ESC was cultured for 8 days solely or with the addition of medroxyprogesterone (MPA) or danazol.

ELISA was done to measure IL-6, IL-8, and TNF-alpha concentrations of the culture media.

Real-time quantitative RT-PCR was done to measure IL-6, IL-8, and TNF-alpha RNA levels in ESC.

ELIGIBILITY:
Inclusion Criteria:

* women with adenomyosis
* at early- to mid-secretory phases

Exclusion Criteria:

* postmenopausal
* malignancy

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45
Dates: Start 2004-07; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Overall Officials: Jehn-Hsiahn Yang, M.D., Principal Investigator — Department of Obstetrics and Gynecology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan